CLINICAL TRIAL: NCT03705533
Title: Single Dose, Full Replicate, Crossover Comparative Bioavailability Study of Telmisartan 80 mg Tablets in Healthy Male and Female Volunteers / Fasting State
Brief Title: Bioequivalence Study of Two Formulations of Telmisartan 80 mg Tablets in Healthy Adult Volunteers Under Fasting State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Algorithme Pharma, An Altasciences Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PTL-P3-923
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Bioequivalence
Keywords: telmisartan; bioequivalence; Micardis
MeSH Terms: interventions — Telmisartan

STUDY DESIGN:
Intervention Model Description: In compliance with full replicate design there are two sequences in the study: ABAB and BABA where A = the test product, B = the reference product (see detailed description of items below).
Who Masked: Outcomes Assessor
Masking Description: *The randomization code will not be available to the personnel of the bioanalytical facility until the bioanalytical tables have been finalized and audited by the Quality Assurance (QA) department. Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence ABAB (Other): Subjects assigned to sequence ABAB will receive a single 80 mg dose of the test product Telmisartan (1 x 80 mg tablet) marked as A in the sequence in Periods 1 and 3 and a single 80 mg dose of the reference product Micardis (1 x 80 mg tablet) marked as B in the sequence in periods 2 and 4. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Telmisartan; Drug: Micardis
- Sequence BABA (Other): Subjects assigned to sequence BABA will receive a single 80 mg dose of the reference product Micardis (1 x 80 mg tablet) marked as B in the sequence in periods 1 and 3 and a single 80 mg dose of the test product Telmisartan (1 x 80 mg tablet) marked as A in the sequence in Periods 2 and 4. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Telmisartan; Drug: Micardis

INTERVENTIONS:
Drug: Telmisartan — Telmisartan is manufactured by Pharmtechnology LLC, Belarus. Each tablet contains 80 mg of telmisartan.
  Other Names: the test product
Drug: Micardis — Micardis is manufactured by Boehringer Ingelheim Ellas AE, Greece. Each tablet contains 80 mg of telmisartan.
  Other Names: the reference product

SUMMARY:
This single center, randomized, single dose, full replicate, crossover comparative laboratory-blinded study will be conducted in healthy male and female volunteers in order to determine the bioequivalence of two different formulations of telmisartan 80 mg tablets after oral administration under fasting conditions.

DETAILED DESCRIPTION:
The study is characterized by single center, randomized, single dose, laboratory-blinded, 4-period, 2-sequence, full replicate crossover design.The objective is to determine the bioequivalence of two different formulations of telmisartan after a single oral dose administration under fasting conditions. The test product is Telmisartan 80 mg tablets manufactured by Pharmtechnology LLC, Belarus. The reference product is Micardis 80 mg tablets manufactured by Boehringer Ingelheim Ellas AE, Greece. The primary study endpoints are the pharmacokinetic parameters Cmax and AUC0-T of telmisartan.

Eligible 26 healthy adult subjects will be randomized to the one of two predetermined sequences: ABAB or BABA where A = the test product, B = the reference product. Clinical part of the study will include 4 periods; in each of them a single 80 mg dose of telmisartan will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast. Wash-out period between treatment administrations will last at least 14 calendar days.

Subjects will be confined to the clinical site from at least 10 hours prior to each drug administration until 24 hours following each drug administration. Subjects will return to the clinical site for the remaining blood samples.

In each study period, 21 blood samples will be collected for pharmacokinetic assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 72 hours after drug administration (0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 postdose) .

Total study duration: up to 74 days (including screening).

Telmisartan plasma concentrations will be measured by a validated bioanalytical method.

Statistical analysis of pharmacokinetic parameters will be based on an ANOVA model. Two-sided 90% confidence interval of the ratio of geometric LSmeans will be obtained from the ln-transformed pharmacokinetic parameters.

Statistical inference of telmisartan will be based on a bioequivalence approach using the following standards:

* average bioequivalence (the ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the test and the reference product for the ln-transformed parameters Cmax and AUC0-T should all be within the 80.00 to 125.00% bioequivalence range);
* scaled-average-bioequivalence (in the event that the Cmax reference-to-reference within-subject CV is greater than 30%, that its test-to-reference geometric LSmeans ratio is within the bioequivalence range of 80.00 125.00% and the average bioequivalence criteria are not met, a scaling approach to the bioequivalence assessment will be used).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy male or female adult volunteer
4. A female volunteer meeting one of the following criteria:

   * (1) Physiological postmenopausal status, defined as the following:

     * absence of menses for at least one year prior to the first study drug administration (not due to amenorrhea secondary to lactation); and
     * Follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at screening; OR
   * (2) Surgical postmenopausal status, defined as the following:

     * bilateral oophorectomy; and
     * absence of menses for at least 90 days prior to the first study drug administration; and
     * FSH levels ≥ 40 mIU/mL at screening; OR
   * (3) Hysterectomy with FSH levels ≥ 40 mIU/mL at screening

   If the postmenopausal volunteer has an FSH of < 40 mIU/mL, but meets the above criteria in either (1), (2) or (3) and all the other inclusion criteria, the volunteer may be included in the study if the estradiol serum level measured at screening is equal to or below 150 pmol/L. In the case of hysterectomy, if FSH and estradiol do not meet the criteria, inclusion of the volunteer will be based on medical judgment.
5. Volunteer aged at least 18 years but not older than 55 years
6. Volunteer with a body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Light-, non- or ex-smoker. A light smoker is defined as someone using 10.0 nicotine units or less per day for at least 90 days prior to the first study drug administration. An ex smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration
8. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

Exclusion Criteria:

1. Females who are pregnant according to the pregnancy test at screening
2. Seated blood pressure below 105/60 mmHg at the screening visit or prior to the first study drug administration
3. History of significant hypersensitivity to telmisartan or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Presence of significant gastrointestinal, liver or kidney disease, or any other condition known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
5. History of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability, including but not limited to cholecystectomy
6. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
7. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
8. History of rare hereditary problems of fructose, galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption
9. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
10. Any clinically significant illness in the 28 days prior to the first study drug administration
11. Use of any prescription drugs (with the exception of hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the volunteer as healthy
12. Any history of tuberculosis
13. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
14. Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests
15. Volunteers who have already been included in a previous group for this clinical study
16. Volunteers who took telmisartan in the 28 days prior to the first study drug administration
17. Volunteers who took an Investigational Product (IP) in the 28 days prior to the first study drug administration
18. Volunteers who donated 50 mL or more of blood in the 28 days prior to the first study drug administration
19. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Cmax of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-T of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration

SECONDARY OUTCOMES:
Tmax of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
TLQC of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Time of last observed quantifiable concentration
AUC0-∞ of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-T + ĈLQC/λZ, where ĈLQC is the predicted concentration at time TLQC
Residual area of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Extrapolated area (i.e. percentage of AUC0-∞ due to extrapolation from TLQC to infinity)
TLIN of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Time point where the log-linear elimination phase begins
λZ of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve
Thalf of telmisartan for the test and the reference products | Time points 0.00 (prior to drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after drug administration
  Terminal elimination half-life, calculated as ln(2)/λZ

OTHER OUTCOMES:
Number of treatment-related adverse events (AE) for the test and the reference products | From the first dosing until 3 days after the collection of the last blood sample of the study
  The safety population will include all subjects who received at least one dose of one of the investigational products. All AEs will be graded as mild, moderate, or severe according to the pre-specified definitions. The qualified investigator will determine the relationship of any AE to the study drug using pre-specified criteria (reasonable possibility or no reasonable possibility). Classification of AEs will be performed by System Organ Class (SOC) and Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA), version 20.1 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Altasciences Company Inc. (doing business as Algorithme Pharma)
Locations (1):
- Algorithme Pharma, An Altasciences Company, Mount Royal, Quebec, Canada